CLINICAL TRIAL: NCT06511544
Title: Repetitive Transcranial Magnetic Stimulation of the Ventromedial Prefrontal Cortex to Target Neural Connectivity and Rumination in Treatment-Resistant Major Depressive Disorder: A Pilot Study
Brief Title: rTMS to Target Neural Connectivity and Rumination in Treatment-Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Susan K. Conroy, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13322; K12TR004415 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Depression, Treatment Resistant
Keywords: transcranial magnetic stimulation; functional magnetic resonance imaging
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active TMS (Experimental): All participants will receive active TMS to the VMPFC for 20 sessions
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — rTMS delivered at 1 Hz for 1800 pulses over 30 minutes for 20 daily sessions, 5 days/week. Treatment will be directed to the ventromedial prefrontal cortex using each participant's structural MRI.

SUMMARY:
The goal of this clinical trial is to learn if Transcranial Magnetic Stimulation (TMS) to part of the brain called the ventromedial prefrontal cortex (VMPFC) can treat a symptom called rumination in adults with major depression that has not responded to at least one medication trial. The main question it aims to answer are:

Does TMS to the VMPFC change brain activity on functional magnetic resonance imaging (fMRI) during a negative self-referential processing task in adults with depression? Does TMS to the VMPFC affect rumination in adults with depression? Researchers will compare brain scans and rumination scores before, during, and immediately after TMS.

Participants will:

Undergo three functional MRI scans Undergo a course of 20 TMS treatments Respond to clinical questionnaires and complete a computer behavioral task

DETAILED DESCRIPTION:
This will be a single-site, pilot, open-label, within-subject design study. 20 participants with treatment-resistant depression, defined as a failure to respond to at least one antidepressant medication trial within a current major depressive episode, will be recruited. Prior to intervention, participants will undergo self-report and clinician-administered assessments (in-person or virtual with both audio and video on using secure health telecommunication method), as well as a fMRI during resting state and a self-referential processing task. The baseline scan will also include a high-resolution structural sequence for neuronavigational purposes. Then, participants will receive 20 daily (5 days/week) sessions of rTMS to the VMPFC along with weekly assessments. Participants will undergo a repeated fMRI scan early in the course of treatment (after session 5) when we would expect neural changes to be evident but prior to any robust overall antidepressant effect, as well as at the end of the rTMS course (after session 20). Scores on the depression and rumination scales will be recorded prior to intervention and weekly thereafter. Contact with subjects will be conducted once via telephone at two weeks after the end of study intervention as an adverse event assessment. In the event that new or persistent adverse events felt to be related to the study intervention occur following the termination of study procedures, subjects may be brought in for further safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar major depressive disorder without psychotic features by the Mini-International Neuropsychiatric Interview (MINI) and confirmed by study psychiatrist
* First depressive episode prior to age 50
* Current moderate to severe depression, Hamilton Depression Rating Scale (HDRS) ≥17)
* Failure to respond to ≥1 antidepressant medication at adequate dose and duration in the current depressive episode; (note: this criterion is designed to be consistent with the original 2008 FDA-labeled indication for TMS in Major Depressive Disorder, that specifies failure to respond to "one prior medication at or above the minimal effective dose and duration in the current episode" (https://www.accessdata.fda.gov/cdrh_docs/pdf8/K083538.pdf). ))
* Off psychotropic medications OR on a stable dose of medication(s) for 6 weeks, and willing to remain on stable medication dosage throughout the study
* Capacity to consent
* Ability to safely receive MRI

Exclusion Criteria:

* Actively/imminently suicidal, Quick Inventory of Depressive Symptomatology (QIDS) item 12 score >2)
* Current depressive episode duration > 5 years
* Presence of clinically significant psychiatric diagnoses other than unipolar, non-psychotic major depression, such as post-traumatic stress disorder (PTSD) or obsessive-compulsive disorder (OCD)
* Evidence of cognitive impairment, Montreal Cognitive Assessment (MOCA) < 23)
* Significant substance use disorder within past 6 months
* New-onset psychotherapy and/or somatic therapy (e.g., light therapy) within 6 weeks of screening
* Prior exposure to any form of TMS
* Have participated in any clinical trial with an investigational drug or device within the past 6 weeks prior to screening
* Failure to respond to Electroconvulsive therapy (ECT)
* Any history of neurosurgery to treat a neurologic or psychiatric disorder (e.g. Vagus nerve stimulation, cortical stimulation, deep brain stimulation, or ablative surgery)
* Unstable medical illness
* Evidence or history of significant neurological disorder, including moderate-severe head trauma, stroke, Parkinson's disease or other movement disorder (except benign essential tremor)
* Epilepsy
* History of seizures (except juvenile febrile seizures or provoked seizures at the PI's discretion) or any condition/concurrent medication that could notably lower seizure threshold
* Pregnancy or planned pregnancy during the study
* Presence of cardiac pacemaker, cochlear implant, or other implanted electronic device
* Any vision problem that will prevent them from seeing the adjectives presented inside the MRI scanner without glasses

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity | Before Transcranial magnetic stimulation (TMS) - immediately following TMS
  Within-network functional connectivity of the default mode network during negative processing
Rumination | Before TMS- immediately following TMS
  Scores on the Ruminative Response Scale (Range 22-88, with higher worse)

SECONDARY OUTCOMES:
Overall Depression Scores | Before TMS- immediately following TMS
  Hamilton Depression Rating Scale (Range 0-52, with higher worse)

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Conroy, MD PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Goodman Hall Neuroscience Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No